CLINICAL TRIAL: NCT05175950
Title: A Placebo-controlled, Randomized, Observer-blinded, Multi-center Study to Assess the Safety, Reactogenicity, and Immunogenicity of Booster Vaccination of A SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510)
Brief Title: Safety, Reactogenicity, and Immunogenicity Study of Heterologous Booster Vaccination of a SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Hee Jin Cheong, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIS_2021_001
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 (Healthy Volunteers)
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Test group 1: primary vaccination completed with ChAdOx1 nCOV-19 (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 1: primary vaccination completed with ChAdOx1 nCOV-19 (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 2: primary vaccination completed with BNT162b2(Pfizer) (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 2: primary vaccination completed with BNT162b2(Pfizer) (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 3: primary vaccination completed with mRNA-1273(Moderna) (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 3: primary vaccination completed with mRNA-1273(Moderna) (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 4: primary vaccination completed with Ad26.COV2.S(Janssen) (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 4: primary vaccination completed with Ad26.COV2.S(Janssen) (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 5: primary vaccination completed with ChAdOx1 nCOV-19(AZ)-BNT162b2(Pfizer) (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 5: primary vaccination completed with ChAdOx1 nCOV-19-BNT162b2 (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 6: primary and 1st booster vaccination completed with mRNA vaccine (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 6: primary and 1st booster vaccination completed with mRNA vaccine (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline
- Test group 7: primary and 1st booster vaccination completed with ≥1 dose of non-mRNA vaccine (Experimental): GBP510 adjuvanted with AS03 (Receptor Binding Domain (RBD) 25μg/dose), 1 dose on Days 0
  Interventions: Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03
- Placebo group 7: primary and 1st booster vaccination completed with ≥1 dose of non-mRNA vaccine (Placebo Comparator): Participants will receive intramuscular (IM) injections of Normal saline on Days 0
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03 — SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) (RBD of SARS-CoV-2 25ug / dose) Adjuvanted with AS03, 1 dose
  Arms: Test group 1: primary vaccination completed with ChAdOx1 nCOV-19; Test group 2: primary vaccination completed with BNT162b2(Pfizer); Test group 3: primary vaccination completed with mRNA-1273(Moderna); Test group 4: primary vaccination completed with Ad26.COV2.S(Janssen); Test group 5: primary vaccination completed with ChAdOx1 nCOV-19(AZ)-BNT162b2(Pfizer); Test group 6: primary and 1st booster vaccination completed with mRNA vaccine; Test group 7: primary and 1st booster vaccination completed with ≥1 dose of non-mRNA vaccine
Other: Normal saline — Normal saline
  Arms: Placebo group 1: primary vaccination completed with ChAdOx1 nCOV-19; Placebo group 2: primary vaccination completed with BNT162b2(Pfizer); Placebo group 3: primary vaccination completed with mRNA-1273(Moderna); Placebo group 4: primary vaccination completed with Ad26.COV2.S(Janssen); Placebo group 5: primary vaccination completed with ChAdOx1 nCOV-19-BNT162b2; Placebo group 6: primary and 1st booster vaccination completed with mRNA vaccine; Placebo group 7: primary and 1st booster vaccination completed with ≥1 dose of non-mRNA vaccine

SUMMARY:
This is randomized, placebo-controlled, observer-blinded, multi-center study to assess safety, reactogenicity and immunogenicity of booster vaccination of a SARS-CoV-2 recombinant protein nanoparticle vaccine (GBP510) adjuvanted with AS03 in adults aged 19 years and older who received a primary series of vaccination or the 1st booster vaccination against COVID-19 approved in Korea.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of booster vaccination of a SARS-CoV-2 recombinant protein nanoparticle vaccine (GBP510).

(Cohort 1~5) A total of approximately 550 adults will be divided into 5 cohorts based on primary series vaccines they received - ChAdOx1 nCOV-19, BNT162b2, mRNA-1273, Ad26.COV2.S and heterologous vaccination with ChAdOx1 nCOV-19 & BNT162b2.

(Cohort 6~7) A total of approximately 220 adults will be divided into 2 cohorts based on primary series & 1st booster vaccines they received -mRNA vaccines (BNT162b2 or mRNA-1273) and at least more than a single dose of non-mRNA vaccines (ChAdOx1 nCOV-19, Ad26.COV2.S, and NVX-CoV2373)

The participants are then randomized at a ratio of 10:1 to either Test Group or Placebo Group. Participants will be subject to follow-up for 12 months after receiving a single booster dose of GBP510 adjuvanted with AS03.

Blood sampling for cell-mediated immunity will be undertaken on approximately 20% of the participants in each cohort, who are selected in advance in consideration of the randomization ratio between Test Group and Placebo Group.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be aged 19 years and older at the time of signing the informed consent.
2. Participants who are healthy or medically stabilized according to medical judgment of the investigator based on medical history, physical examination and clinical laboratory tests, etc.
3. Participants who are able to attend all scheduled visits and comply with all study procedures.
4. (Cohort 1~5) Participants who received a primary series of COVID-19 vaccination approved for use in Korea by MFDS and at least 12~24 weeks have passed with no additional COVID-19 vaccination.
5. (Cohort 6~7) Participants who received a primary series of COVID-19 vaccination and the 1st booster vaccination at least 16 weeks ago through a homologous or heterologous vaccination with mRNA vaccines (BNT162b2 (Pfizer) and mRNA-1273 (Moderna)) only or at least more than a single dose of non-mRNA vaccines (ChAdOx1 nCOV-19 (AZ), Ad26.COV2.S (Janssen), and NVX-CoV2373 (Novavax)).
6. Female participants of childbearing potential must agree to be heterosexually inactive, or agree to use at least one acceptable method of contraception from at least 4 weeks prior to the study vaccination (booster vaccination) to 12 weeks after the study vaccination.
7. Female participants with a negative urine or serum pregnancy test at screening (However, female participants who are surgically sterile or postmenopausal with amenorrhea for at least 12 months shall be excluded.
8. Participants who give signed informed consent which include compliance with the requirements and restrictions listed in the informed consent form and in the protocol.

Exclusion Criteria:

1. Any clinically significant respiratory symptoms (e.g. cough, sore throat), febrile illness (temperature >38°C), or acute illness within 72 hours prior to the study vaccination (A prospective participant should not be included until 72 hours after the condition has resolved).
2. History of virologically-confirmed COVID-19, SARS or MERS disease.
3. History of confirmed SARS-CoV-2 infection within three months before screening.
4. History of congenital or acquired immunodeficiency or autoimmune disease.
5. History of bleeding disorder including thrombocytopenia which is judged by the investigator as a contraindication for intramuscular vaccination.
6. History of hypersensitivity and severe allergic reaction (e.g. anaphylaxis, Guillain-Barre syndrome) to any components of the study intervention.
7. History of malignancy within 1 year prior to the study vaccination (Except for a participant judged by the investigator to have a low recurrence risk.)
8. Any other clinically significant conditions such as uncontrollable chronic or acute diseases which, in the opinion of the investigator, might cause a health threat to the participant or interfere with the clinical trial procedures or interpretation of the study results.
9. Any other conditions which might interfere with the evaluation of the study objectives (e.g. alcohol or drug abuse, neurologic or psychiatric conditions).
10. Female participants who are pregnant or breastfeeding.
11. History of drug administration other than COVID-19 vaccination intended to treat or prevent COVID-19.
12. History or planned other vaccination within 4 weeks prior to the study vaccination through 28 days after the study vaccination (except for influenza vaccination, which may be received at least 2 weeks prior to the study vaccination).
13. Receipt of immunoglobulins, whole blood or blood products within 12 weeks prior to the study vaccination.
14. Use of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy for at least 2 consecutive weeks within 12 weeks prior to the study vaccination or long-term systemic corticosteroid therapy (e.g. ≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) (However, the use of topical and nasal glucocorticoids will be permitted.)
15. History of participation in another clinical study within 4 weeks prior to the study vaccination or planned participation in another clinical study during this study period.
16. Investigators, study staff who are directly involved in the conduct of this study or supervised by the investigator, or their family members.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Comparative GMT (Geometric Mean Titer) of neutralizing antibody to SARS-CoV-2 between the Test Group and Placebo Group, measured by wild-type virus neutralization assay at 2 weeks post heterologous booster vaccination | Through Day 365 post last vaccination
GMT (Geometric Mean Titer) of SARS-CoV-2 RBD-binding antibody measured by ECLIA at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
GMFR (Geometric Mean Fold Rise) of SARS-CoV-2 RBD-binding antibody from baseline measured by ECLIA at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
Percentage of participants with ≥4-fold rise from baseline in SARS-CoV-2 RBD-binding antibody measured by ECLIA at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
GMT (Geometric Mean Titer) of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
GMFR (Geometric Mean Fold Rise) of neutralizing antibody to SARS-CoV-2 from baseline measured by wild-type virus neutralization assay at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
Percentage of participants with ≥4-fold rise from baseline in neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay at each time point post heterologous booster vaccination | Through Day 365 post last vaccination
(Only applicable to CMI analysis set) Cell-mediated immunity assessment using IFN-γ ELISpot at each time point post heterologous booster vaccination | Through Day 365 post last vaccination

SECONDARY OUTCOMES:
Occurrence of immediate systemic reactions | in 30 minutes post heterologous booster vaccination
Occurrence of solicited local AEs during 7 days post heterologous booster vaccination | Through 7 days post-vaccination
Occurrence of solicited systemic AEs during 7 days post heterologous booster vaccination | Through 7 days post-vaccination
Occurrence of unsolicited AEs during 28 days post heterologous booster vaccination | Through 28 days post-vaccination
Occurrence of SAEs, MAAEs and AESIs during the study period | Through Day 0 to Day 365 post vaccination

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Korea University Ansan Hospital, Ansan
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Hallym University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju